CLINICAL TRIAL: NCT05627557
Title: A Phase III, International, Multicenter, Randomised Open Label Study to Evaluate the Efficacy and Safety of Obinutuzumab Versus MMF in Patients With Childhood Onset Idiopathic Nephrotic Syndrome
Brief Title: A Study to Evaluate the Efficacy and Safety of Obinutuzumab Versus MMF in Participants With Childhood Onset Idiopathic Nephrotic Syndrome
Acronym: INShore
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WA43380; 2022-000369-42 (EudraCT Number); 2023-505140-19-00 (Other: EU CT Number)
Record Dates: First submitted 2022-11-04; First posted 2022-11-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Childhood Idiopathic Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — obinutuzumab; Prednisone; Methylprednisolone; Acetaminophen; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obinutuzumab (Group A) (Experimental): Participants in Group A will receive obinutuzumab 1000 milligrams (mg) (or 20 mg/ kilogram [kg] for participants <45 kg) administered by intravenous (IV) infusion on Days 1, 15, 168 (Week 24), and 182 (Week 26).
  Interventions: Drug: Obinutuzumab; Drug: Prednisone; Drug: Methylprednisolone; Drug: Acetaminophen/ Paracetamol; Drug: Diphenhydramine Hydrochloride
- MMF (Group B) (Active Comparator): Participants in Group B will receive oral MMF 600 mg/m^2 twice a day (BID) (target 1200 mg/m2/day in divided doses, maximum 2 g/day) to Week 52.
  Interventions: Drug: MMF; Drug: Prednisone

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab will be administered as per schedule specified in the respective arm.
  Arms: Obinutuzumab (Group A)
Drug: MMF — MMF will be administered as per schedule specified in the respective arm.
  Arms: MMF (Group B)
Drug: Prednisone — Participants taking prednisone or equivalent at randomization will follow a guided tapering schedule to reach the goal of 0mg/day by Weeks 4-6 (and no later than Week 8 following randomization and continue without prednisone through Week 52.
  Other Names: Non-Investigational Medicinal Product
Drug: Methylprednisolone — Methylprednisolone 80 mg (or 1.5 mg/kg if </=45 kg) IV will be administered as premedication prior to infusions.
  Other Names: Non-Investigational Medicinal Product
  Arms: Obinutuzumab (Group A)
Drug: Acetaminophen/ Paracetamol — Acetaminophen 15 mg/kg (maximum dose 1000 mg) will be administered PO as premedication prior to infusions.
  Other Names: Non-Investigational Medicinal Product
  Arms: Obinutuzumab (Group A)
Drug: Diphenhydramine Hydrochloride — Diphenhydramine HCl 0.5-1 mg/kg (maximum dose 50 mg) will be administered PO or IV as premedication prior to infusions.
  Other Names: Non-Investigational Medicinal Product
  Arms: Obinutuzumab (Group A)

SUMMARY:
This open-label, randomized multicenter study is to assess the efficacy, safety, and pharmacokinetics (PK)/pharmacodynamics (PD) of obinutuzumab compared with mycophenolate mofetil (MMF) in children and young adults (aged >= 2-25 years) with frequently relapsing nephrotic syndrome (FRNS) or steroid-dependent nephrotic syndrome (SDNS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of frequently relapsing nephrotic syndrome (FRNS) or steroid dependent nephrotic syndrome (SDNS) before the age of 18 years
* Must be in complete remission defined by the absence of edema, UPCR <= 0.2 g/g at screening and have three consecutive daily urine dipstick readings of trace or negative for protein within the week prior to randomization
* Must have had at least one relapse in the 6 months prior to screening, after discontinuation of or while receiving oral corticosteroids and/or immunosuppressive therapy to prevent relapses
* Participants having received cyclophosphamide in the 6 months prior to randomization must have experienced at least 1 relapse subsequent to cyclophosphamide discontinuation
* Estimated glomerular filtration rate (eGFR) within normal range for age
* For females of childbearing potential: participants who agree to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraception, during the treatment period and for 18 months after the final dose of obinutuzumab and for 6 weeks after the final dose of MMF
* For males: participants who agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agree to refrain from donating sperm during the treatment period and for 90 days after the final dose of MMF

Exclusion Criteria:

* Secondary nephrotic syndrome
* History of steroid resistant nephrotic syndrome
* History of genetic defects known to directly cause nephrotic syndrome
* Treatment with other immunosuppressive medications to prevent relapse, other than MMF or oral corticosteroids within 2 months prior to randomization
* Pregnancy or breastfeeding or intending to become pregnant during the study or within 18 months after the final dose of obinutuzumab, or within 6 weeks after the final dose of MMF
* Females of childbearing potential, including those who have had a tubal ligation, must have a negative serum pregnancy test result within 28 days prior to initiation of study treatment and a negative urine pregnancy test at Day 1, prior to randomization
* History of organ or bone marrow transplant
* Participation in another therapeutic trial within 30 days of enrollment or 5 half-lives of the investigational drug
* Intolerance or contraindication to study therapies
* Participants demonstrating prior treatment failure to MMF as defined by two or more relapses in any 6-month period of time while receiving MMF for at least a 6-month duration
* Participants in the judgment of the investigator likely to require systemic corticosteroids for reasons other than idiopathic nephrotic syndrome during the study
* Active infection of any kind or any major episode of infection requiring hospitalization or treatment with IV anti-infective medications within 4 weeks prior to screening, or completion of oral anti-infectives within 2 weeks prior to randomization
* History of or currently active primary or secondary immunodeficiency, including known history of human immunodeficiency virus (HIV) infection and other severe Immunodeficiency blood disorders
* History of progressive multifocal leukoencephalopathy
* History of or current cancer, including solid tumors, hematological malignancies, and carcinoma in situ within the past 5 years
* Major surgery requiring hospitalization during the 4 weeks prior to screening or during screening
* High risk for clinically significant bleeding or any condition requiring plasmapheresis, intravenous immunoglobulin, or acute blood product transfusions
* Evidence of any significant or uncontrolled concomitant disease that, in the investigator's judgment, would preclude participant's participation, including but not limited to nervous system, respiratory, cardiac, hepatic, endocrine, malignant, or gastrointestinal disorders
* Currently active alcohol or drug abuse or history of alcohol or drug abuse

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2026-09-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Sustained Complete Remission at 1 year | At Week 52

SECONDARY OUTCOMES:
Overall Relapse-free Survival (RFS) | At Week 52
Probability of RFS at Week 52 | At Week 52
Cumulative Corticosteroid Dose | At Week 52
Number of Relapses | At Week 52
Percentage of Participants Experiencing Edema Associated Relapse | At Week 52
Percentage of Participants with Sustained Complete Remission | Week 52 to Week 76
  This outcome measure will be assessed at primary analysis
Mean Change in "General Fatigue" Domain of Pediatric Quality of Life Inventory (PedsQL) Multidimensional Fatigue Scale Total Score | Baseline to Week 52
Mean Change in "Physical Functioning" Domain of PedsQL Quality of Life Inventory | Baseline to Week 52
Mean Change in Cure Glomerulonephropathy (CureGN) Edema Scale | Baseline to Week 52
Percentage of Participants with Adverse Events (AEs) | Baseline to Week 52
Serum Concentrations of Obinutuzumab | At Days 1, 15 28, 84, 168, 182, 224, 364, and at Early Study Discontinuation Visit (unscheduled visit at the time of discontinuation from study, any time between Day 1 and Day 364)
Percentage of Participants Achieving B Cell Depletion Highly Sensitive Flow Cytometry (HSFC) | At Days 1, 15, 28, 84, 168, 224, 364, and at Early Study Discontinuation Visit (unscheduled visit at the time of discontinuation from study, any time between Day 1 and Day 364)
Total Peripheral B Cell and B Cell Subsets (e.g., Memory B Cells) Counts and Change from Baseline | At Days 1, 15, 28, 84, 168, 224, 364, and at Early Study Discontinuation Visit (unscheduled visit at the time of discontinuation from study, any time between Day 1 and Day 364)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- United States (10):
  - Lucile Packard Children's Hospital - Stanford, Palo Alto, California
  - Memorial Healthcare System, Hollywood, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Children's Healthcare of Atlanta Center for Advanced Pediatrics, Atlanta, Georgia
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Levine Children's Hospital, Charlotte, North Carolina
  - University of Utah - Primary Children's Hospital - PPDS, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
- UZ Gent, Ghent, Belgium
- Brazil (3):
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto Hospital de Base - PPDS, São José do Rio Preto, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
- China (6):
  - Peking University First Hospital, Beijing
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The children's hospital , Zhejiang university school of medicine, Hangzhou
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Xi'an Children's Hospital, Xi'an
  - Henan Children's Hospital Zhengzhou Children's Hospital, Zhengzhou
- France (4):
  - Chu Toulouse, Toulouse, Haute-Garonne
  - Hopital Femme Mere Enfants, Bron
  - Hopital Henri Mondor, Créteil
  - Hopital Robert Debre, Paris
- Italy (2):
  - Istituto G Gaslini Ospedale Pediatrico IRCCS - INCIPIT - PIN, Genoa, Liguria
  - Ospedale Infantile Regina Margherita - INCIPIT - PIN, Turin, Piedmont
- Japan (9):
  - Tokyo Metropolitan Children's Medical Center, Fuchu-Shi
  - Hokkaido University Hospital, Hokkaido
  - Hyogo prefectural Kobe Children's Hospital, Hyogoken
  - Kobe University Hospital, Kobe
  - Shiga University Of Medical Science Hospital, Ōtsu
  - Kitasato University Hospital, Sagamihara-Shi
  - Dokkyo Medical University Hospital, Shimotsuga-Gun
  - National Center for Child Health and Development, Tokyo
  - Yokohama City University Medical Center, Yokohama
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Dzieciecy Szpital Kliniczny UCK WUM, Warsaw
- Spain (2):
  - Hospital Sant Joan de Deu - PIN, Espluges de Llobregat, Barcelona
  - Hospital Universitario Cruces, Barakaldo, Vizcaya

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526
- [Derived] Dossier C, Bonneric S, Baudouin V, Kwon T, Prim B, Cambier A, Couderc A, Moreau C, Deschenes G, Hogan J. Obinutuzumab in Frequently Relapsing and Steroid-Dependent Nephrotic Syndrome in Children. Clin J Am Soc Nephrol. 2023 Dec 1;18(12):1555-1562. doi: 10.2215/CJN.0000000000000288. Epub 2023 Sep 6. PMID 37678236